CLINICAL TRIAL: NCT01551069
Title: A Randomized, Double Blind, Baseline Controlled Study Using Placebo as Reference for Assessing the Efficacy and Safety of Hydroxychloroquine Sulfate in Patients With Systemic Lupus Erythematosus or Cutaneous Lupus Erythematosus in the Presence of Active Lupus Erythematosus Specific Skin Lesion
Brief Title: Multicenter Study Assessing the Efficacy & Safety of Hydroxychloroquine Sulfate in Patients With Systemic Lupus Erythematosus or Cutaneous Lupus Erythematosus With Active Lupus Erythematosus Specific Skin Lesion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC12368; U1111-1126-8072 (Other: UTN)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Cutaneous Lupus Erythematosus-Systemic Lupus Erythematosus
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCQ (Active Comparator): HCQ 200~400mg, once daily, oral administration
  Interventions: Drug: hydroxychloroquine (Z0188)
- Placebo (Other): HCQ-placebo, once daily, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydroxychloroquine (Z0188) — Pharmaceutical form:tablet
  Route of administration: oral
  Other Names: Plaquenil®
  Arms: HCQ
Drug: Placebo — Pharmaceutical form:tablet
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

- To investigate the efficacy on skin manifestation of 16 weeks treatment of once daily regimen of hydroxychloroquine sulphate (HCQ) in patients with cutaneous lupus erythematosus (CLE) and systemic lupus erythematosus (SLE) with active skin manifestation (CLASI [Cutaneous Lupus Erythematosus Disease Area and Severity Index] activity score is ≥4) concomitant treatment with or without corticosteroid.

Secondary Objectives:

* To evaluate the efficacy on skin manifestation and the safety of 16 weeks treatment of once daily regiment of HCQ versus placebo as the reference group in patients with CLE and SLE with active skin manifestation (CLASI activity score is ≥4) concomitant treatment with or without corticosteroid.
* To investigate the safety of 16 weeks treatment of once daily regiment of HCQ in patients with CLE and SLE with active skin manifestation concomitant treatment with or without corticosteroid.
* To investigate the safety and efficacy of 52 weeks long-term treatment of once daily regimen of HCQ in patients with CLE and SLE - To investigate the influence of the dose reduction of corticosteroid on CLE and SLE patients treated with HCQ concomitant with corticosteroid
* To investigate efficacy of once daily regimen of HCQ on systemic symptoms, musculoskeletal symptoms and immunological parameters in SLE patients.

DETAILED DESCRIPTION:
Total 59 weeks (screening;4 weeks, treatment;52 weeks, Follow-up; 3 weeks)

ELIGIBILITY:
Inclusion criteria :

* Patients diagnosed as cutaneous lupus erythematosus (CLE)

Exclusion criteria:

* Patients receiving corticosteroid more than 15mg/day of the equivalent dose of prednisolone.
* Patients whose CLASI activity scores were less than 4 point at the initiation of Screening (Visit 1) and Day1 (Visit 2) (evaluated by a dermatology specialist).
* Patients whose fluctuations of CLASI activity scores were ≥20% between Visit 1 and Visit 2 (evaluated by a dermatology specialist). The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
A change in CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index) activity score | from baseline (at visit 2) to 16 weeks treatment (at visit 6)

SECONDARY OUTCOMES:
A change in CLASI activity score | from baseline (at visit 2) to 52 weeks treatment (at visit 15)
BILAG (British Isles Lupus Assessment Group) index to be conducted in patients complicated with SLE | 7 timepoints during 52 weeks
RAPID 3 (Routine assessment of patient index data 3) to be conducted in patients complicated with SLE : daily life activity, pain associated with the original disease, patient's severity related to the original disease | 7 timepoints during 52 weeks
QOL related to skin manifestations (skindex-29) | 4 timepoints during 52 weeks
Dose reduction of concomitant corticosteroid | From 16 weeks to 55 weeks after the initiation of the treatment
Global assessment by investigator (skin and other) | 3 timepoints during 52 weeks
Global assessment by patient (skin) | 3 timepoints during 52 weeks
Immunological parameters | up to maximum of 13 timepoints during 52 weeks
Number of patients with serious adverse events / adverse events | up to a maximum of 59 weeks
Ophthalmologic examination (visual acuity examination, slit-lamp examination, funduscopic examination, visual field examination and color vision examination) | 14 timepoints during 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- Japan (22):
  - Investigational Site Number 392017, Bunkyō City
  - Investigational Site Number 392022, Bunkyō City
  - Investigational Site Number 392011, Chuo-Ku, Kumamoto-Shi
  - Investigational Site Number 392003, Chūōku
  - Investigational Site Number 392001, Fuchu-Shi
  - Investigational Site Number 392008, Iruma-Gun
  - Investigational Site Number 392009, Iruma-Gun
  - Investigational Site Number 392005, Itabashi-Ku
  - Investigational Site Number 392014, Kamogawa
  - Investigational Site Number 392019, Kanazawa
  - Investigational Site Number 392007, Kitakyushu
  - Investigational Site Number 392020, Maebashi
  - Investigational Site Number 392012, Nagasaki
  - Investigational Site Number 392010, Nagoya
  - Investigational Site Number 392013, Nakagami-Gun
  - Investigational Site Number 392006, Sagamihara-Shi
  - Investigational Site Number 392018, Sagamihara-Shi
  - Investigational Site Number 392002, Shinjuku-Ku
  - Investigational Site Number 392023, Tomigusuku-Shi
  - Investigational Site Number 392021, Uruma
  - Investigational Site Number 392004, Wakayama
  - Investigational Site Number 392016, Yokohama

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Yokogawa N, Eto H, Tanikawa A, Ikeda T, Yamamoto K, Takahashi T, Mizukami H, Sato T, Yokota N, Furukawa F. Effects of Hydroxychloroquine in Patients With Cutaneous Lupus Erythematosus: A Multicenter, Double-Blind, Randomized, Parallel-Group Trial. Arthritis Rheumatol. 2017 Apr;69(4):791-799. doi: 10.1002/art.40018. PMID 27992698